CLINICAL TRIAL: NCT02519751
Title: Total Body Skeletal Muscle Mass Estimation by Creatine (Methyl-d3) Dilution in Athletes
Brief Title: New Method Using Deuterium Labelled Creatine to Measure Total Body Skeletal Muscle Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202600
Record Dates: First submitted 2015-07-23; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Sports Nutritional Sciences
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- D3 Creatine followed by creatine supplementation (Experimental): Every participant will be orally administered with 60mg of D3 Creatine in a fasted state in a non-gelatin capsule. Creatine supplemented throughout the study will be administered in the following doses-0.03, 0.035, 0.04, 0.045 g.kg.Lean mass/day, increasing on weekly basis. Final dose of 0.05 g.kg.Lean mass/day is then maintained throughout the study.
  Interventions: Dietary Supplement: D3 Creatine; Dietary Supplement: Creatine

INTERVENTIONS:
Dietary Supplement: D3 Creatine — One dose of D3 Creatine (60mg capsule) given orally on Day 1
Dietary Supplement: Creatine — Participants will consume an individual dosed level of creatine, based on their estimated muscle mass in doses of 0.03, 0.035, 0.04, 0.045 g.kg.Lean mass/day, increasing on a weekly basis. Final dose of 0.05 g.kg.Lean mass/day is then maintained throughout the study.

SUMMARY:
Creatine (methyl-d3) dilution (D3-creatine) is a novel technique for the estimation of muscle mass. The method uses a dose of deuterium-labelled creatine to determine total skeletal muscle mass via estimation of total body creatine pool size.The aim of this study is to compare estimates of total body skeletal muscle mass by D3-creatine dilution method and whole body Magnetic Resonance Imaging (MRI) in an athletic population.

ELIGIBILITY:
Inclusion Criteria:

* Trained and competing elite canoe athletes will be recruited, who represent Great Britain Canoeing

Exclusion Criteria:

* Pregnant and lactating women
* Intolerance or hypersensitivity to Creatine supplementation
* Athletes with disabilities which affect their total body muscle mass
* If creatine was taken in a supplemented form, rather than dietary intake, more regularly than once a week within 6-weeks of assessment commencing
* Contraindication to an MRI scan

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Correlation between muscle mass obtained by MRI method and D3-Creatine method | Upto 3 months
  MRI scan of the participants will be done at Day 1 and end of study (i.e.Day 90).D3-Creatine capsule will be given orally at Day 1 and urine samples collected at 0-4h and 4-24h every day from Day 1 to Day 4.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Brentford, United Kingdom